CLINICAL TRIAL: NCT02780037
Title: To Motivate Elderly to Move: Focus on Prevention or Promotion?
Brief Title: To Motivate Elderly to Move
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: S58680
Record Dates: First submitted 2016-02-23; First posted 2016-05-23 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2016-02

CONDITIONS: Geriatric Disorder

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Prevention (Experimental): Regulatory frame: prevention
  Interventions: Behavioral: Regulatory frame: prevention
- Promotion (Experimental): Regulatory frame: promotion
  Interventions: Behavioral: Regulatory frame: promotion
- Neutral (Sham Comparator): Regulatory frame: not implied
  Interventions: Behavioral: Regulatory frame: not implied

INTERVENTIONS:
Behavioral: Regulatory frame: prevention — Exercise program presented as preventing deterioration.
  Arms: Prevention
Behavioral: Regulatory frame: promotion — Exercise program presented as promoting improvement.
  Arms: Promotion
Behavioral: Regulatory frame: not implied — Exercise program presented without implied consequences.
  Arms: Neutral

SUMMARY:
This study examines the short- and long-term-effects of different repeated frames in which an exercise program is offered on behavior (i.e., frequency of exercise) and motivation (i.e., autonomous/controlled) in older people (65+). The frames are manipulated experimentally as either prevention focused (e.g., to prevent worse health), promotion focused (e.g., to gain better health) or neutral (control condition).

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age

Exclusion Criteria:

* severe mental/physical problems

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 111 (Actual)
Dates: Start 2016-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Behavior at long term: exercise frequency during third week | third week
  self-reported no exercise sessions

SECONDARY OUTCOMES:
Change in controlled motivation over long term: end week 3 - baseline | 3 weeks
  baseline, end week 3 (BREQ-2 questionnaire)
Change in autonomous motivation over long term: end week 3 - baseline | 3 weeks
  baseline, end week 3 (BREQ-2 questionnaire)
Change in controlled motivation over short term: end week 1 - baseline | 1 week
  baseline, end week 1 (BREQ-2 questionnaire)
Change in autonomous motivation over short term: end week 1 - baseline | 1 week
  baseline, end week 1 (BREQ-2 questionnaire)
Behavior at short term: exercise frequency during first week | first week
  self-reported no exercise sessions

OTHER OUTCOMES:
Functionality: sit to stand/sit: flexion, extension, stand and sit duration (time) | week 1/week 2/week 3
  (Dynaport)
Functionality: sit to stand/sit: angular velocity flexion and extension (degrees/sec) | week 1/week 2/week 3
  (Dynaport)
Functionality: sit to stand/sit: range flexion and extension (degrees) | week 1/week 2/week 3
  (Dynaport)
Functionality: SPPB (Short Physical Performance Battery) score | week 1/week 2/week 3
  (Dynaport)
Functionality: SPPB balance score | week 1/week 2/week 3
  (Dynaport)
Functionality: SPPB gait speed score | week 1/week 2/week 3
  (Dynaport)
Functionality: SPPB chair stand score | week 1/week 2/week 3
  (Dynaport)
Functionality: sway acceleration (mG) | week 1/week 2/week 3
  (Dynaport)
Functionality: sway velocity (mm/sec) | week 1/week 2/week 3
  (Dynaport)
Functionality: sway path (mm/sec) | week 1/week 2/week 3
  (Dynaport)
Functionality: sway normalized area (mm²/sec) | week 1/week 2/week 3
  (Dynaport)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Kinesiology, Heverlee, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vanroy J, Seghers J, van Uffelen J, Boen F. Can a framed intervention motivate older adults in assisted living facilities to exercise? BMC Geriatr. 2019 Feb 18;19(1):46. doi: 10.1186/s12877-019-1060-z. PMID 30777017